CLINICAL TRIAL: NCT06479005
Title: Early Detection of Clinical Deterioration Using an Integrated Remote Monitoring System in Lung Cancer Patients Receiving Cytotoxic Chemotherapy.
Brief Title: ETERNALS: Remote Monitoring in Lung Cancer Patients
Acronym: ETERNALS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z2023080
Record Dates: First submitted 2024-06-12; First posted 2024-06-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Remote Monitoring; Mobile Health; Chemotherapy Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Monocentric prospective interventional feasibility study
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional feasibility study arm (Experimental): Patients will receive a wearable device to monitor vital parameters continuously from the first round of chemo until the last cycle (approx 15 weeks).
  Interventions: Device: Oura Ring

INTERVENTIONS:
Device: Oura Ring — The Oura ring will remotely monitor the patients vitals at home continuously

SUMMARY:
The primary objective of this project is to determine the feasibility of an integrated remote monitoring system in the routine care of lung cancer patients receiving cytotoxic chemotherapy.

DETAILED DESCRIPTION:
Lung cancer is a highly prevalent malignant tumor with 5.563 new cases in Belgium in 20201. Up to 70% of patients present with locally advanced or metastatic disease at diagnosis 1. Most of these patients require systemic therapy including cytotoxic chemotherapy as part of their treatment plan. The mortality rate in this patient population remains high due to the aggressive nature of the disease, but also due to treatment related toxicities such as dehydration, infection, and anemia, resulting in emergency department (ED) visits and rehospitalizations. Routine administration of highly effective anti-emetics and the use of granulocyte colony-stimulating growth factors greatly reduced the complication rate in these patients 2, 3. Also, remote symptom monitoring using a web-based tool to which patients can self-report their toxicities (i.e., patient-reported outcomes; PROs) had a marked impact on reducing ED visits and increasing overall survival in the patient-reported outcome (PRO) group 4-6. Despite these successes there is still a large proportion of lung cancer patients for whom weekly self-reports are not feasible. More specific: low socio-economic status, elderly patients and social isolation are associated with low compliance 7, 8. The latter lung cancer patient subgroup is at the highest risk of under-detection when presenting with treatment- or disease-related toxicity. The investigators hypothesize that implementation of an integrated remote monitoring system tracking heart rate, heart rate variability, body temperature, respiration rate, nocturnal oxygen saturation, sleep tracking and daily activity level via an unobtrusive wearable device is more performant and less burdensome compared to other self-reporting methods (e.g., PROs). The primary aim of this project is to set up and implement an integrated remote monitoring system in the routine care of lung cancer patients receiving cytotoxic chemotherapy, in which the remote monitoring is enabled via an unobtrusive wearable device. Via this innovative implementation the investigators believe that patient care can be drastically improved due to the earlier detection of deterioration (i.e., less rehospitalizations and ED visits), especially for those high-risk frail patients.

ELIGIBILITY:
Inclusion Criteria:-

* Patient must be in the possession of a phone
* Diagnosis of Stage IV lung cancer patients treated with cytotoxic chemotherapy
* Older than 18 years of age

Exclusion Criteria:

* Life expectancy of less than 6 weeks
* Not able to understand the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time interval | 18 months
  Determining the time interval between clinical deterioration detected by the integrated remote monitoring system and the first contact with the care team (i.e., in current clinical practice the patient suffering from chemotherapy-associated symptoms self-reports at the ED)
Compliance | 18 months
  Patient compliance in using the integrated remote monitoring system which will be determined via: number of missed measurements, number of telephonic/physical contact moments related to the technology

SECONDARY OUTCOMES:
System Usability scale to assess usability and acceptability of the remote monitoring system | 18 months
  Acceptability and usability of the integrated remote monitoring system by both the patient and the healthcare specialists. This will be assessed using the following questionnaire: System Usability scale (SUS). The scale varies from 1-5, corresponding with 1 being strongly disagree and 5 strongly agree. Depending on the question, the score can be found either positive/negative.
mobile Health App Usability Questionnaire to assess usability & acceptability of the remote monitoring system | 18 months
  Acceptability and usability of the integrated remote monitoring system by both the Acceptability and usability of the integrated remote monitoring system by both the patient and the healthcare specialists. This will be assessed using the following questionnaire: mobile Health App Usability Questionnaire (MAUQ). The scale varies from 1-7, with 1 corresponding to 'disagree' and 7 corresponding to 'agree'. Depending on the question, the score can be found either positive/negative.
Number of ED visits | 18 months
  Determine the number of ED visits retrospectively, including the disease- and therapy related/induced complications (retrospective sub-study)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Criel, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06479005/Prot_SAP_000.pdf